CLINICAL TRIAL: NCT01437228
Title: Does Preoperative Vaginal Preparation With Povidone-iodine Before Cesarean Delivery Reduce the Risk of Endometritis?
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Erzincan Military Hospital (Other)
Responsible Party: Principal Investigator, Kemal GUNGORDUK, Mardin Women and Children Hospital, Erzincan Military Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: gungorduk13
Record Dates: First submitted 2011-09-06; First posted 2011-09-20 (Estimated); Last update posted 2011-11-17 (Estimated); Status verified 2011-11

CONDITIONS: Postpartum Endometritis

ARMS (2):
- povidone iodine (Other): 30-second vaginal scrub with povidone- iodine solution.
  Interventions: Drug: povidone- iodine solution.
- CONTROL (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: povidone- iodine solution. — %10 Polivinilpirolidon iyot (Polividon- iyot
  Other Names: BATTICON Solüsyon. Adeka
  Arms: povidone iodine
Drug: placebo — NO İNTERVENTİON
  Other Names: NO İNTERVENTİON
  Arms: CONTROL

SUMMARY:
Cesarean delivery rates are increasing in Turkey and a major component of this increase is cesarean on demand. Although data on the rate of cesarean delivery in Turkey is limited, a national study reported a rate of 23.8%. Infectious morbidity, consisting primarily of endomyometritis and wound infection, remains a leading cause of postoperative complications. Estimates of postcesarean infection rates range from 7% to 20%, depending on demographic and obstetric variables. Infection following cesarean delivery results in not only increased hospital stay but also increases the cost of care. Strategies to minimize postoperative infectious and other morbidities have included modifications of surgical technique, changing of gloves, methods of placental delivery, cervical dilatation during cesarean delivery, and altering the uterine position during repair of the uterine incision. Despite these interventions, endometritis is still major problem after cesarean delivery.

Endometritis appears to result from ascending vaginal flora bacteria, with anaerobes playing an important role. The microbes endogenous to the vagina change throughout the course of pregnancy and parturition. Larsen and Galask noted that anaerobic species located in the vagina increase dramatically by the third postpartum day. In many cases, the surgeon's hand, reaching below the infant's head or presenting part, is in direct contact with the vagina. Vaginal bacterial flora have been cultured from the delivering surgeon's glove in 79% (95% confidence interval [CI] 58%, 100%) of cesareans that follow labor. In these cases, vaginal flora are delivered directly to the uterus, abdominal cavity, and the abdominal incision. Vaginal preparation has been shown to decrease the quantitative load of vaginal microorganisms as well as to remove certain species of bacteria.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 38 weeks estimated gestational age and required cesarean section.

Exclusion Criteria:

* Highly emergent cesarean
* Allergy to povidone iodine
* Chorioamnionitis on admission
* Fever on admission

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 668 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
rate of postpartum endometritis | 6 weeks
  Endometritis was defined here as body temperature greater than 38.5C with concomitant foul-smelling discharge or abnormally tender uterus on bimanual examination

SECONDARY OUTCOMES:
morbidity | two days
  Infectious morbidity was documented using established clinical criteria. Febrile morbidity was defined as a persistent fever of at least 38C for at least 24 hours after surgery and not associated with lower abdominal or pelvic tenderness and no signs of infection elsewhere.

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Etfal Hospital, Istanbul, Sisli, Turkey (Türkiye)

REFERENCES:
- [Derived] Haas DM, Morgan S, Contreras K, Kimball S. Vaginal preparation with antiseptic solution before cesarean section for preventing postoperative infections. Cochrane Database Syst Rev. 2020 Apr 26;4(4):CD007892. doi: 10.1002/14651858.CD007892.pub7. PMID 32335895